CLINICAL TRIAL: NCT06652230
Title: Assessment of Treatment Efficacy Using Smile Arc Marginal Ridge Approach Versus MBT Chart Method for Bracket Positioning: A Randomized Clinical Trial
Brief Title: Assessment of Treatment Efficacy Using Smile Arc Marginal Ridge Approach Versus MBT Chart Method for Bracket Positioning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Medhat Mostafa Kamal Abdelaziz, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42/7/24
Record Dates: First submitted 2024-10-11; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Class I Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Smile Arc Marginal Ridge Approach (SAMRA) (Experimental)
  Interventions: Other: Smile Arc Marginal Ridge Approach (SAMRA)
- MBT Chart Method (Active Comparator)
  Interventions: Other: MBT Chart Method

INTERVENTIONS:
Other: Smile Arc Marginal Ridge Approach (SAMRA) — Smile Arc Marginal Ridge Approach (SAMRA) is a new orthodontic bonding technique proposed by Dr. Dalia El Bokle where she stated that it provides more accurate orthodontic results and less time and effort needed during finished. No randomized clinical trials are done on this new approach yet so our study is the first one to test it. 0.018-inch MBT brackets will be used in our study.
  Arms: Smile Arc Marginal Ridge Approach (SAMRA)
Other: MBT Chart Method — For our comparator group MBT Chart Method will be used. Using charts during orthodontic bonding procedures is considered the gold standard. 0.018-inch brackets will be used.
  Arms: MBT Chart Method

SUMMARY:
The goal of this randomized clinical trial is to evaluate the effect of Smile Arc Marginal Ridge Approach (SAMRA) versus MBT chart method for bracket positioning on orthodontic treatment results.

The main questions it aims to answer are:

Is there a difference in orthodontic treatment results between smile arc marginal ridge approach (SAMRA) and MBT chart method for bracket positioning?

Does SAMRA provide more accurate orthodontic results and reduce the number of archwire bendings and brackets repositioning needed during finishing?

The investigators will compare Smile Arc Marginal Ridge Approach (SAMRA) with MBT Chart Method (gold standard) to see if SAMRA provides more accurate orthodontic results and reduce the need for archwire bendings and brackets repositioning during finishing.

Participants will:

* Undergo orthodontic treatment and divided into two groups, Group A (SAMRA) and Group B (MBT Chart Method).
* 0.018-inch MBT brackets will be used in both groups.
* Follow ups every 1 month will take place to change the archwires after becoming passive.
* After leveling and alignment is completed, orthodontic treatment results, number of archwire bendings and brackets repositioning needed will be determined to see which type of intervention is better or if both provide similar results.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patients aged 11-30 years old.
* Mild or moderate crowding not requiring tooth extraction.
* Full permanent dentition including fully erupted 7s not necessarily 8s.
* Good oral hygiene.
* Skeletal and dentoalveolar class I malocclusion.

Exclusion Criteria:

* Systemic disease potentially affecting the study outcome.
* Cleft lip and palate/syndromic patients.
* Any signs or symptoms of temporomandibular disorders (TMD).
* Previous orthodontic treatment.
* Pregnant females.
* Chronic use of medications.

Ages: 11 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Orthodontic treatment results | 6 months
  Orthodontic treatment results will be assessed according to the American Board of Orthodontics Objective Grading System (ABO-OGS) using the ABO measuring gauge.

SECONDARY OUTCOMES:
Number of additional archwire bending and bracket repositioning needed | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided